CLINICAL TRIAL: NCT05787899
Title: Efficacy of the Hepatitis B Vaccination Post Hypothermia for Hypoxic Ischemic Encephalopathy
Brief Title: Hypothermia's Effect on Hepatitis B Vaccination
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Florian Capobianco, Resident, Medical University of South Carolina
Other Study IDs: Pro00126670
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Hepatitis B Vaccination; Hypothermia, Newborn
Keywords: Hypoxic Ischemic Encephalopathy; Hepatitis B vaccination
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypothermia Protocol
  Interventions: Other: Hypothermia Protocol

INTERVENTIONS:
Other: Hypothermia Protocol — Subject's who will be treated with the hypothermia protocol for Hypoxic Ischemic Encephalopathy as standard of care.

SUMMARY:
The purpose of the research is to determine if the Hepatitis B vaccine after birth provides enough protection after cooling for Hypoxic Ischemic Encephalopathy (HIE). To do this, Hepatitis B titers (blood sample) would be taken before, during, and after administering of the Hepatitis B vaccine series to measure efficacy of the vaccine.

DETAILED DESCRIPTION:
Despite the current research on Hypoxic Ischemic Encephalopathy (HIE), and the known effects of hypothermia on acute immune response, the effect of the hypothermia protocol for HIE on the efficacy of the Hepatitis B vaccine is still unknown. We plan to measure anti-hepatitis B surface antibodies at intervals prior, during, and after the primary Hepatitis B vaccine schedule for individuals with HIE to see if there is any effect on efficacy due to the Hypothermia protocol.

ELIGIBILITY:
Inclusion Criteria:

* > 34 weeks' gestation at birth as measured by best obstetrical estimates
* > 1500 grams birth weight
* Clinical signs of asphyxia or documented periods of hypoxic ischemia with no cyanotic cardiac malformations and no known congenital infections.
* Documented period of hypoxic ischemia:
* Venous Cord gas pH < 7.0 or initial newborn blood gas pH < 7.1
* Base deficit > 13 on venous cord gas or initial newborn blood gas
* Apgar score < 5 at 10 minutes
* Prolonged, sustained fetal bradycardia (HR <80) for > 15 minutes in utero by doppler or fetal heart rate monitoring
* Need for continued resuscitation after 5 minutes (bag-valve mask ventilation with/or without chest compressions) due to the absence of respiratory effort
* Documented postnatal oxygen saturation < 70% or PaO2 < 35 for > 20 minutes by 2 ABGs, not due to cyanotic heart disease, accompanied by hypotension (mean BP< 35), cardiac arrest with chest compressions, or hemorrhage (requiring 20cc/kg volume replacement)
* Parental willingness for infant to receive Hepatitis B vaccine.

Exclusion Criteria:

- Positive maternal Hepatitis B status during pregnancy

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hypothermia protocol is only approved for HIE in newborn infants and thus only newborn infants will be subjects in this study. We enroll every neonate who meets entry criteria or is referred for HIE to our institutions regardless of race and gender.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Determine efficacy of the Hepatitis B vaccine in individuals who are treated with routine care of Hypothermia for Hypoxic Ischemic Encephalopathy | 18 months
  Response to vaccine will be measured by the previously researched protective level of anti-hepatitis B surface antibodies of ≥ 10 mIU/ml. We hypothesize that hypothermia to 33-33.5oC for 72h in near-term and term infants with Hypoxic Ischemic Encephalopathy will decrease the infant's immune response to the primary Hepatitis B vaccine series.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No